CLINICAL TRIAL: NCT03229291
Title: A Phase 1, Single-Center, Randomized, Single-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of SM04755 Following Topical Administration to Healthy Subjects
Brief Title: A Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of SM04755 Following Topical Administration to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM04755-TOP-01
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Tendinopathy
Keywords: SM04755; topical; Samumed; Wnt inhibitor
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose (Experimental): Topical SM04755 solution (15 mg/mL) applied once per day for 14 days
  Interventions: Drug: SM04755
- Mid Dose (Experimental): Topical SM04755 solution (45 mg/mL) applied once per day for 14 days
  Interventions: Drug: SM04755
- High Dose (Experimental): Topical SM04755 solution (90 mg/mL) applied once per day for 14 days
  Interventions: Drug: SM04755
- Vehicle (Placebo Comparator): Vehicle solution applied once per day for 14 days
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SM04755 — SM04755 is a small molecule inhibitor of the Wnt pathway.
  Arms: High Dose; Low Dose; Mid Dose
Drug: Vehicle — Same formulation as topical SM04755 solution, without SM04755 included.
  Arms: Vehicle

SUMMARY:
This study is a single-center, randomized, single-blind, placebo-controlled, multiple ascending dose study of SM04755 solution applied topically once daily for 14 days to intact skin overlying the inner thigh of healthy subjects at an estimated body surface area (BSA) of 80 cm^2. Dosing cohorts will consist of 8 subjects who will be randomized 3:1 (SM04755:placebo).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18 to 30 kg/m^2 at study start
* Subject must have read and understood the informed consent form, and must have signed it prior to any study-related procedure being performed
* Willingness to comply with all scheduled study visits, laboratory tests, contraception requirements and other study procedures
* Appropriate skin characteristics at site of application (inner thigh) (for example, consistent pigmentation, no tattoos, no scarring or noted injury, no varicose veins or structural repair)
* Willing to avoid extensive sun exposure, phototherapy, or use of a tanning salon for the duration of the study

Exclusion Criteria:

* Women who are pregnant or lactating
* Women of childbearing potential who are sexually active and are not willing to use a highly effective method of birth control during the study period that includes double barrier, intrauterine device (IUD), or hormonal contraceptive combined with single barrier, or abstinence
* Males who are sexually active and not willing to use a condom, and have a partner who is capable of becoming pregnant, if neither has had surgery to become sterilized, and/or who are not willing to use double barrier or whose partner is not using a highly effective method of birth control (e.g., IUD or hormonal contraception combined with single barrier).
* History of, or current, skin disease (for example, psoriasis, atopic dermatitis, seborrheic dermatitis, and skin cancer)
* History of, or current, skin damage at the treatment site (inner thigh) (for example, cuts, abrasion, sunburn, sun-damage, or scarring)
* Phototherapy or use of a tanning salon 2 weeks prior to study start until end of the study (Day 28)
* History of, or current, allergy to investigational product/placebo ingredients
* Known allergy to adhesive tape
* Current evidence of malignancy or history of malignancy within the last 5 years prior to study start; prior history of in situ cancer or basal or squamous cell skin cancer, completely excised, is allowed
* Treatment with an investigational product within 12 weeks prior to study start; the last date of participation in the trial, not the last date of receipt of investigational product, must be at least 12 weeks prior to study start
* Use of any prescription or nonprescription drugs [except birth control or hormone replacement therapy (HRT)], topical skin treatments on the application site (inner thigh), vitamins, grapefruit/grapefruit juice, or dietary or herbal supplements within 14 days prior to study start
* Blood donation of ≥ 1 pint (473 mL) within 56 days prior to study start or unwilling to refrain from blood donation for the duration of the study
* Plasma or platelet donation within 14 days prior to study start or unwilling to refrain from plasma or platelet donation for the duration of the study
* Unwilling to refrain from sperm donation for the duration of the study and until 90 days after dose administration
* Prior or current latent or active tuberculosis (TB) or nontuberculous mycobacteria infection.
* Evidence of active infection or illness involving fever within 7 days prior to study start
* Occurrence of serious illness requiring hospitalization within 6 months prior to study start
* Regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months prior to study start
* Use of tobacco- or nicotine-containing products (cigarettes, pipe, cigar, chewing tobacco or nicotine gum, lozenges or patches) within 30 days prior to study start
* A history of abuse of prescription or illicit drugs within 6 months prior to study start
* Marijuana use within 28 days prior to study start
* Previous treatment with SM04755
* Subjects who have a current or pending disability claim, workers' compensation, or litigation(s) that may compromise response to treatment
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative site, or are directly affiliated with the study at the investigative site
* Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-06-11 (Actual); Study Completion 2017-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Day 28
  Incidence and severity of AEs events during the treatment and observation periods of the study
Incidence of clinical laboratory abnormalities | Day 28
  Incidence and severity of clinical laboratory measurements that are outside the normal range
Change in vital signs: blood pressure | Baseline and Day 28
  Change from baseline in blood pressure
Change in vital signs: temperature | Baseline and Day 28
  Change from baseline in temperature
Change in vital signs: respiratory rate | Baseline and Day 28
  Change from baseline in respiratory rate
Change in vital signs: pulse rate | Baseline and Day 28
  Change from baseline in pulse rate
Change in electrocardiogram (ECG) parameters | Baseline and Day 28
  Change from baseline in 12-lead ECG parameters
Plasma pharmacokinetics (PK): Cmax | Day 1
  Maximum plasma concentration (Cmax) estimate for SM04755 following first dose
Plasma pharmacokinetics (PK):tmax | Day 1
  Time to Cmax estimate for SM04755 following first dose
Plasma pharmacokinetics (PK): AUC | Day 1
  Area under the plasma concentration-time curve (AUC) estimate for SM04755 following first dose
Plasma pharmacokinetics (PK):half-life | Day 1
  Plasma terminal phase half-life estimate for SM04755 following first dose
Plasma pharmacokinetics (PK):Cmax | Day 14
  Maximum plasma concentration (Cmax) estimate for SM04755 following last dose
Plasma pharmacokinetics (PK):tmax | Day 14
  Time to Cmax estimate for SM04755 following last dose
Plasma pharmacokinetics (PK): AUC | Day 14
  AUC estimate for SM04755 following last dose
Plasma pharmacokinetics (PK):half-life | Day 14
  Plasma terminal phase half-life estimate for SM04755 following last dose
Change in skin score assessment: erythema | Baseline and Day 28
  Change from baseline in erythema skin score assessment
Change in skin score assessment: scaling | Baseline and Day 28
  Change from baseline in scaling skin score assessment
Change in skin score assessment: pruritus/itching | Baseline and Day 28
  Change from baseline in pruritus/itching skin score assessment
Change in skin score assessment: burning/stinging | Baseline and Day 28
  Change from baseline in burning/stinging skin score assessment

SECONDARY OUTCOMES:
Incidence of AEs relative to exposure | Day 28
  Incidence and severity of AEs relative to measured plasma exposure to SM04755

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (1):
- Research Site, Tempe, Arizona, United States